CLINICAL TRIAL: NCT06390982
Title: A Single-arm, Multicenter, Phase II Clinical Study of Chemoradiotherapy Followed by Tislelizumab Combined With Chemotherapy for Organ Preservation in Resectable Low Rectal Cancer：the RELIEVE-01 Study
Brief Title: Organ Preservation With Tislelizumab and Total Neoadjuvant Therapy in Patients With Low Rectal Cancer: RELIEVE -01 Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Shanghai Changzheng Hospital (Other); Huadong Hospital (Other); RenJi Hospital (Other); Hebei Medical University Fourth Hospital (Other); First Hospital of China Medical University (Other); Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Xu jianmin, Chief Physician, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-2011-IIT
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: RECTAL NEOPLASMS; Rectal Cancer
Keywords: tislelizumab; low rectal cancer; organ preservation; watch and wait; TNT
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; tislelizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tislelizumab (Experimental): CRT followed by 4 cycles of tislelizumab plus CAPOX and clinical response assessment:
  participants with CR (cCR+ pCR confirmed by local resection of ncCR): another 4 cycles of tislelizumab plus CAPOX and 9 cycles of tislelizumab, then watch and wait.
  participants with non-CR: underwent TME
  Interventions: Radiation: Radiotherapy; Drug: Tislelizumab; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Radiation: Radiotherapy — 45-50.4Gy in 25-28 fractions to the pelvis on Days 1-5 every week.
Drug: Tislelizumab — 200 mg IV on Day 1 of each 21-day cycle.
Drug: Capecitabine — Capecitabine 1000 mg/m2 orally twice daily (bid) on Day 1 to 14 of each 21-day cycle in CAPOX regimen
Drug: Oxaliplatin — 130 mg/m2 IV on Day 1 of each 21-day cycle in CAPOX regimen
Drug: Capecitabine — 825 mg/m2 orally twice daily (bid) 5 days/week during radiotherapy.

SUMMARY:
This is an open-label, multi-center, single-arm clinical study. All patients received concurrent chemoradiation therapy (CRT) followed by 4 cycles of tislelizumab combined with CAPOX, then underwent clinical response assessment. Patients who achieved CR (cCR+ pCR confirmed by local resection of ncCR) continue tislelizumab combined with CAPOX for another 4 cycles and tislelizumab for 9 cycles, then Watch and Wait. Patients who did not achieved CR underwent total mesorectal excision (TME).

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent, understand and comply with the requirements and evaluation schedule
2. ≥18, ≤75 years old
3. Histologically confirmed rectal adenocarcinoma
4. immunohistochemistry confirmed pMMR (positive for MLH1, MSH2, MSH6 and PMS2), or PCR /NGS confirmed MSI-L or MSS
5. The distance from the lower edge of the tumor to the anal verge is ≤5 cm through colonoscopy, digital anal examination or MRI
6. clinical stage cT1-3N1M0 or cT2-3N0M0 (the 8th UICC/AJCC; T and N is evaluated by MRI)
7. Resectable primary tumor assessed by the Investigator
8. Have not received any anti-tumor treatment for rectal cancer
9. ECOG PS ≤ 1
10. Adequate organ function
11. Female subjects with the ability to become pregnant must have a serum pregnancy test with a negative result within 72 hours before the first dose, and be willing to use highly effective contraceptive methods during the trial and 120 days after the last dose. Male subjects whose partners are women of childbearing potential should be surgically sterilized or agree to use a highly effective method of contraception during the trial and for 120 days after the last dose.

Exclusion Criteria:

1. Histologically confirmed poorly differentiated/undifferentiated adenocarcinoma, mucinous adenocarcinoma and signet ring cell carcinoma
2. Have received any treatments for rectal cancer, or evidence of distant metastasis
3. Presence of following high risk factors assessed by MRI: MRF +, EMVI+, cN2, Positive lateral lymph nodes, T3d
4. Presence or in high risk of obstruction, perforation or bleeding;
5. Not suitable for long-course radiotherapy
6. Cannot tolerate surgery
7. ≥2 colorectal cancer lesions at the same time
8. Contraindications for MRI examination
9. Other malignant tumors in the past or at the same time
10. Have an active autoimmune disease requiring systemic therapy within the past 2 years
11. HIV infection
12. Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers (HBV DNA > 500 IU/mL) or active HCV carriers with detectable HCV RNA;
13. Hypersensitivity to any ingredient of tislelizumab, capecitabine, and oxaliplatin or to any component of the container
14. Other conditions judged by the researcher that do not meet the enrollment requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 46 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Complete Response rate (CR rate) | From first dose up to 12 months, approximately
  defined as the proportion of participants with clinical complete response(cCR) or near clinical complete response (ncCR) who achieved local resection confirmed pCR determined by the investigators after CRT and 4 cycles of CAPOX plus tislelizumab.

SECONDARY OUTCOMES:
1/2/3 year organ-preservation rate | From first dose of radiotherapy up to 36 months, approximately
  defined as the proportion of participants who survived and did not underwent TME in 1/2/3 year (in the CR set and full analysis set respectively)
1/2/3 year EFS rate | From first dose of radiotherapy up to 36 months, approximately
  defined as the proportion of participants who did not develop local recurrence, distant metastasis, new invasive primary lesions of colorectal cancer, or death in 1/2/3 year (in the CR set, non-CR set and full analysis set respectively)
1/2/3 year OS rate | From first dose of radiotherapy up to 36 months, approximately
  defined as the proportion of participants who survived in 1/2/3 year (in the full analysis set)
Percentage of Participants With Adverse Events | From first dose of radiotherapy up to 36 months, approximately
  Percentage of Participants With adverse events (AEs) , immune-related adverse events(irAE) and serious adverse events (SAEs) per the National Cancer Institute CommonTerminology Criteria for Adverse Events (NCI CTCAE) Version 5.0

IPD SHARING:
Plan to Share IPD: No